CLINICAL TRIAL: NCT06708325
Title: Effects of Resistance Exercise-based Physical Activity Programme on Physical and Psychological Factors in Inactive Adults
Brief Title: Effect of Resistance Exercise on Physical and Psychological Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monira Aldhahi (Other)
Collaborators: Namik Kemal University (Other)
Responsible Party: Sponsor-Investigator, Monira Aldhahi, Professor, Princess Nourah Bint Abdulrahman University
Organization: Princess Nourah Bint Abdulrahman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.135.06.21; Tekirdağ Namık Kemal Universit (Other: Tekirdağ Namık Kemal University)
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Physically Inactive
Keywords: Strength; balance; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants and outcome assessors, the data analysts were masked to group assignment throughout the study. The data analysts were not present during the exercise sessions or assessments and did not have access to information that could potentially reveal whether data belonged to the exercise or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The 12-week resistance training program consisted of three supervised sessions per week, each lasting approximately 55-60 minutes. Sessions were structured as follows: 5-7 minute dynamic warm-up, 35-40 minutes of resistance training, and 4-5 minutes of stretching for active recovery. Participants were paired based on similar strength fitness levels and progressed according to the principle of periodized progressive overload.
  Interventions: Other: Resistance Training Program
- control group (No Intervention): did not participate in any structured exercise program during the 12-week study period. The participants were asked to maintain their usual lifestyle habits.

INTERVENTIONS:
Other: Resistance Training Program — The 12-week resistance training program consisted of three supervised sessions per week, each lasting approximately 55-60 minutes. Sessions were structured as follows: 5-7 minute dynamic warm-up, 35-40 minutes of resistance training, and 4-5 minutes of stretching for active recovery.Participants were paired based on similar strength fitness levels and progressed according to the principle of periodized progressive overload. Training was delivered using a circuit protocol with 2-3 sets per exercise. The initial 4-week phase included 2 sets per exercise, with 8-20 repetitions and 1-2 minutes rest between sets. .The program incorporated functional exercises targeting the lower extremities, core, and upper extremities, utilizing equipment such as resistance bands, medicine balls, jump ropes, dumbbells, bars, and stability balls. Participants performed exercises in a circuit sequence, with the intensity, number of sets, and repetitions
  Arms: Exercise group

SUMMARY:
Physical inactivity is a key risk factor for cardiovascular and metabolic disorders, negatively affecting emotional well-being by increasing psychological distress and reducing mental health. This study aimed to evaluate the impact of a resistance-based physical activity program on physical and psychological outcomes in physically inactive adults.

DETAILED DESCRIPTION:
Background/Objectives: Sedentary behavior is a prevalent risk factor contributing to the development and progression of cardiovascular and metabolic diseases. Additionally, physical inactivity has been linked to diminished emotional well-being, characterized by elevated levels of psychological distress and compromised mental health. The present study was designed to investigate the effects of a resistance-focused physical activity intervention on both physical and psychological health outcomes in adults with chronically low levels of physical activity. A randomized controlled trial design was employed. The participant comprised 32 adults (mean age = 46.61 ± 7.33 years) included in the study. These individuals were randomly allocated to either a resistance exercise group (EG, n = 15) or a control group (CG, n = 17). Comprehensive assessments were conducted at baseline and following the 12-week intervention. These assessments included evaluations of muscle strength (knee flexors, knee extensors, ankle dorsiflexors, plantar flexors, and core isometric strength), static and dynamic balance, proprioception, and functional movement capacity (as measured by the Functional Movement Screen (FMS)). Participants' psychological states were quantified using the Depression, Anxiety, and Stress Scale-21 (DASS-21). The EG participated in a supervised resistance training program 3 days per week for 12 weeks, with each session lasting approximately 55-60 minutes. Conversely, the CG did not engage in any structured exercise program and were advised to maintain their customary lifestyle habits throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40-60 years
* Physically independent
* Not having cardiac, orthopedic, or musculoskeletal dysfunctions
* Not participating in regular physical activity more than once a week for the last 5 months before the beginning of the study

Exclusion Criteria:

* Chronic ankle instability
* Lower extremity musculoskeletal injury in the previous 6 months
* Undergoing hormonal replacement therapy
* Having uncontrolled diabetes
* Having uncontrolled hypertension
* Histroy of cardiovascular disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Depression | From enrollment to the end of treatment at 12 weeks
  The Depression, Anxiety, Stress Scale-21 (DASS-21) is a widely used self-report tool designed to measure depression, anxiety, and stress levels in participants. It consists of 21 items divided into three subscales:
  * Depression (e.g., feelings of sadness, lack of motivation)
  * Anxiety (e.g., nervousness, fearfulness)
  * Stress (e.g., tension, irritability)
  Each item is scored on a 4-point Likert scale, with the following options:
  1. 0 = Did not apply to me at all
  2. 1 = Applied to me to some degree, or some of the time
  3. 2 = Applied to me to a considerable degree, or a good part of the time
  4. 3 = Applied to me very much, or most of the time
  For each subscale, the scores range from 0 to 42 after adjustment.
Functional Movement Screen Test Protocol | From enrollment to the end of treatment at 12 weeks
  a standardized assessment tool designed to evaluate fundamental movement patterns, identify asymmetries and weaknesses, and predict injury risk. The FMS consists of 7 movements: deep squat, hurdle step, in-line lunge, shoulder mobility, active straight leg raise, trunk stability push-up, and rotational stability.Each movement is scored on a 0-3 scale, with 3 indicating optimal performance. The maximum total score is 21.
Balance | From enrollment to the end of treatment at 12 weeks
  Balance was assessed using the Sensbalance MiniBoard (Sensamove®, Utrecht, The Netherlands), a movable platform that provides an interactive challenge to balance control. Participants performed two tasks, each completed twice and held for 30 seconds
Strength tests | From enrollment to the end of treatment at 12 weeks
  Lafayette Manual Muscle Test System (Model 01165) was used to determine isometric muscle strength. The Lafayette Manual Muscle Tester (MMT) system is an ergonomic handheld device used to objectively measure muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Ustaömer, Principal Investigator — Namik Kemal University
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Medicine, Tekirdağ Namık Kemal University, Tekirdağ, Turkey,, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study investigators plan to disseminate the results of this trial through publication in peer-reviewed scientific journals and presentation at relevant conferences. While the investigators are committed to transparency and data sharing, individual participant data (IPD) may not be shared due to the potential risk of identifying participants despite anonymization efforts. Given the specific nature of the interventions and assessments, there is a possibility that participant identities could be inadvertently disclosed.